CLINICAL TRIAL: NCT06882473
Title: A Clinical Study of Pelvic Concurrent Chemoradiotherapy Combined with CT-guided Intracavitary Brachytherapy with Adaptive Simultaneous Dose Escalation for Locally Advanced Cervical Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 797-02
Record Dates: First submitted 2025-02-07; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Cervical Cancer
MeSH Terms: interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment group (Experimental): External beam radiation therapy: The patients are irradiated with 6MV X-rays at 1.8Gy per fraction, 5 fractions per week, with a total dose of 45-50.4Gy in 25-28 fractions for 5-6 weeks.
  Brachytherapy: CT-guided 192Ir high dose rate brachytherapy is used, twice a week, on the same day as external beam radiation therapy, 6Gy per fraction, a total dose of 30Gy. The total radiotherapy dose shouldn't be less than 85Gy EQD2. The overall treatment time ≤ 45 days.
  Chemotherapy: Cisplatin 40 mg/m2, d1, i.v. weekly. Six cycles of concurrent chemotherapy should be completed. Treatment continued until disease progression, unacceptable toxic effects happened, or a decision by the investigator and/or patient to discontinue treatment.
  Interventions: Other: Brachytherapy and CT-guided online adaptive external beam pelvic radiotherapy are delivered on the same day

INTERVENTIONS:
Other: Brachytherapy and CT-guided online adaptive external beam pelvic radiotherapy are delivered on the same day — Brachytherapy and CT-guided online adaptive external beam pelvic radiotherapy are delivered on the same day.

SUMMARY:
The standard treatment for locally advanced cervical cancer is cisplatin-based concurrent chemoradiotherapy with external beam radiotherapy (EBRT) and Brachytherapy (BT). overall treatment time (OTT) has been found to be an important predictor of treatment response. Some studies have shown that the acceleration of tumor cell regeneration during the extension of radiotherapy leads to poor local control. Prolonging the overall treatment time of cervical cancer radiotherapy for more than 8 weeks leads to an increase in pelvic local control failure. Therefore, shortening OTT has great potential benefits from both clinical efficacy and social benefits. Shortening OTT in radical cervical cancer radiotherapy includes hypofractionated EBRT and shortening the interval between BT and EBRT. However, further shortening OTT may lead to an increase in acute and late toxicity. Adaptive radiotherapy (ART) strategies systematically monitor variations in target and neighbouring structures to inform treatment-plan modification during radiotherapy. The application of image-guided adaptive brachytherapy (IGABT) has clearly demonstrated the advantages of this approach in the treatment of cervical cancer. Previous studies have shown that the implementation of IGABT can achieve personalized treatment, dose increase, improve clinical efficacy, reduce normal tissue toxicity and side effects, and strengthen international standardized quality control. In this study, online adaptive pelvic EBRT combined with IGABT based on uRT-linac was performed under online CT guidance.

The aim of this study is to evaluate the safety and efficacy of pelvic concurrent chemoradiotherapy combined with CT-guided intracavitary brachytherapy with adaptive simultaneous dose escalation in locally advanced cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent;
2. Age :18 to 75 years old;
3. Histologically or cytologically confirmed cervical cancer;
4. According to the International Federation of Gynecology and Obstetrics (FIGO 2018) stage IB3, IIA2, IIB, III, IV (local advanced), and had not received treatment before enrollment;
5. Measurable lesions according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1;
6. ECOG physical performance score 0-2;
7. Expected survival time >= 3 months;
8. LVEF >= 55%;
9. Bone marrow function: neutrophil >= 1.5×109/L, platelet ≥ 100×109/L, white blood cell 4.0-10.0×109/L, hemoglobin >= 90 g/L;
10. Liver and kidney function: serum creatinine <= 1.5 times upper limit of normal; AST and ALT≤2.5 times upper limit of normal (ULN) or <= 5 times ULN in the presence of liver metastasis; Total bilirubin <=1.5 times upper limit of normal, or <= 2.5 times upper limit of normal if the patient has Gilbert's syndrome;
11. Subjects of childbearing age must agree to use effective contraception during the trial, and women of childbearing age must have a negative serum or urine pregnancy test;
12. Non-lactating patients;

Exclusion Criteria:

1. Patients with prior abdominal or pelvic radiotherapy;
2. being mentally ill and unable to cooperate with treatment;
3. Serious uncontrolled medical diseases, such as serious internal medical diseases, including severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, uncontrolled infection, active peptic ulcer, etc.;
4. Unable to tolerate cisplatin chemotherapy;
5. receiving other experimental drugs or participating in clinical trials for other anticancer treatment purposes within 30 days before the first radiotherapy;
6. Severe infection within 4 weeks before study treatment, including but not limited to infectious complications requiring hospitalization, bacteremia, or severe pneumonia;
7. Human immunodeficiency virus (HIV) -positive persons;
8. HBsAg positive and HBV-DNA titer >= 1×10^3 IU/mL; Participants were eligible for inclusion if they were HBsAg positive and had a peripheral blood HBV-DNA level of < 1×10^3 IU/mL, and if the investigator considered the participant to be in a stable phase of chronic hepatitis B without increasing the risk to the participant.
9. Hepatitis C virus (HCV) antibody positive or human immunodeficiency virus (HIV) antibody positive and HCV RNA test positive;
10. Patients judged by the investigator to be ineligible for the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
the nature of adverse events | The time frame extends from the initiation of radiotherapy to 24 months after the completion of radiotherapy
  the nature of adverse events is assessd by RTOG/EORTC radiation toxicity grading
the frequency of adverse events | The time frame extends from the initiation of radiotherapy to 24 months after the completion of radiotherapy

SECONDARY OUTCOMES:
objective response rate | The time frame extends from the initiation of radiotherapy to 12 months after the completion of radiotherapy
tumor control rate | The time frame extends from the initiation of radiotherapy to 24 months after the completion of radiotherapy
local progression-free survival time | The time frame extends from the initiation of radiotherapy until the first recorded local recurrence, with an initial assessment period of 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Jiang, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No